CLINICAL TRIAL: NCT05131997
Title: A Randomized, Double-blind, Active-controlled, Multicenter Phase 3 Trial to Evaluate the Efficacy and Safety of Administrated AD-221 and AD-221A in Patients With Primary Hypercholesterolemia
Brief Title: A Study to Evaluate the Efficacy and Safety of AD-221 and AD-221A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD-221P3
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Primary Hypercholesterolemia
MeSH Terms: interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AD-221 (Experimental): AD-221, Placebo of AD-221A, AD-221B and AD-221C
  Interventions: Drug: AD-221
- AD-221A (Experimental): AD-221A, Placebo of AD-221, AD-221B and AD-221C
  Interventions: Drug: AD-221A
- AD-221B (Active Comparator): AD-221B, Placebo of AD-221, AD-221A and AD-221C
  Interventions: Drug: AD-221B
- AD-221C (Active Comparator): AD-221C, Placebo of AD-221, AD-221A and AD-221B
  Interventions: Drug: AD-221C

INTERVENTIONS:
Drug: AD-221 — PO, Once daily(QD), 8 weeks
  Arms: AD-221
Drug: AD-221A — PO, Once daily(QD), 8 weeks
  Arms: AD-221A
Drug: AD-221B — PO, Once daily(QD), 8 weeks
  Other Names: Ezetimibe
  Arms: AD-221B
Drug: AD-221C — PO, Once daily(QD), 8 weeks
  Other Names: Atorvastatin
  Arms: AD-221C

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AD-221 and AD-221A

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of AD-221 and AD-221A in patients with primary hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subjects with primary hypercholesterolemia

Exclusion Criteria:

* Patient with secondary dyslipidemia
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Low density lipoprotein cholesterol (LDL-C) | Baseline, Week 8
  LDL-C change at Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hak Lee, M.D., Ph.D, Principal Investigator — Yonsei University Hospital
Locations (1):
- Yonsei University Hospital, Seoul, Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No